CLINICAL TRIAL: NCT04934774
Title: Non-gene Edited Anti-CD7 CAR T Cells for Relapsed/Refractory T Cell Malignances
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCAR Bio Therapeutics Ltd. (Industry); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG177-001
Record Dates: First submitted 2021-02-27; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Acute Lymphoblastic Lymphoma; T-cell Non-Hodgkin Lymphoma
Keywords: Anti-CD7 CAR; CD7CAR; T cell leukoma/lymphoma; T-ALL; T-cell acute lymphoblastic leukemia; T-cell acute lymphoblastic lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD7 CAR T cells (Experimental): anti-CD7 CAR T cells Dose escalation phase: anti-CD7 CAR T cells transduced with a lentiviral vector to express CD7 chimeric receptor domain on T cells with an escalation approach, 1 e6 to 5 e6 CAR-T cells/kg.
  Interventions: Biological: CD7 CAR T cells

INTERVENTIONS:
Biological: CD7 CAR T cells — Non-gene edited anti-CD7 CAR T cells administered to patients, will be either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of non-gene edited anti-CD7 CAR (also called anti-CD7 CAR) T cells in patients with relapsed and/or refractory T cell lymphoma or leukemia

DETAILED DESCRIPTION:
Anti-CD7 CAR is a chimeric antigen receptor immunotherapy treatment designed to treat leukemia/lymphoma expressing CD7 antigen. T-cell acute lymphoblastic leukemia, T-acute lymphoblastic lymphoma and T-cell non-Hodgkin lymphoma are a subset of leukemias and lymphomas that are positive for the surface protein CD7. The purpose of this study is to evaluate the efficacy and safety of anti-CD7 CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent; Patients volunteer to participate in the research
2. Diagnosis is mainly based on the World Health Organization (WHO) 2008
3. Patients have exhausted standard therapeutic options
4. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 1 weeks
5. Female must be not pregnant during the study

Exclusion Criteria:

1. Patients declining to consent for treatment
2. Prior solid organ transplantation
3. Potentially curative therapy including chemotherapy or hematopoietic cell transplant
4. Any drug used for GVHD must be stopped >1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | The first 28 days after infusion
  Number of participants with dose limiting toxicity (DLT) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Type of dose-limiting toxicity (DLT) | The first 28 days after infusion
  Type of dose-limiting toxicity (DLT)
Adverse event by severity | 2 years
  Number of participants with adverse event by severity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Overall response rate of ant-CD7 CAR | 1 year
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CR1), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS)
Overall survival | 1 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, Principal Investigator — Peking University Shenzhen Hospital, China
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No